CLINICAL TRIAL: NCT01091948
Title: GlideScope Video Laryngoscope vs Fiberoptic Intubation
Brief Title: GlideScope Video Laryngoscope Versus Fiberoptic Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 08-079
Record Dates: First submitted 2010-03-09; First posted 2010-03-24 (Estimated); Results first posted 2016-12-20 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-10

CONDITIONS: Oral Intubation
Keywords: elective general surgery; orotracheal intubation; Patients would be eligible for inclusion if they were at least 18 years old and scheduled for elective surgery requiring orotracheal intubation.
MeSH Terms: interventions — Intubation; Optical Fibers; Laryngoscopes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fiberoptic Intubation (Active Comparator): Subjects will be intubated with the Fiberoptic laryngoscope.
  Interventions: Device: Intubation with Fiberoptic laryngoscope
- GlideScope® Video Laryngoscope (Active Comparator): Subjects will be intubated with the GlideScope® Video Laryngoscope.
  Interventions: Device: GlideScope® Video Laryngoscope

INTERVENTIONS:
Device: Intubation with Fiberoptic laryngoscope — Subjects will be intubated with the Fiberoptic laryngoscope.
  Other Names: Fiberoptic; laryngoscope
  Arms: Fiberoptic Intubation
Device: GlideScope® Video Laryngoscope — Patients will be intubated with the GlideScope® Video Laryngoscope.
  Other Names: GlideScope®; Video Laryngoscope
  Arms: GlideScope® Video Laryngoscope

SUMMARY:
Following informed consent, patients will be randomly assigned to oral fiberoptic intubation or to oral intubation using the GlideScope Video Laryngoscope. Following the induction of general anesthesia a sealed envelope would be opened to reveal the technique to be used. A stop watch will be started at the beginning of the procedure. At the completion of intubation the stop watch will be stopped and the time recorded along with other data. Based on a sample size estimation process, it is the investigators plan to study fifty patients. The two techniques will be compared in terms of the average time needed to place the endotracheal tube and studied using a two-sided T-Test with a significance level of 0.05. To ensure comparability between the two methods, all intubators will be required to have at experienced at least 10 uses of the GlideScope and 10 uses with fiberoptic intubation.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* scheduled for elective surgery requiring orotracheal intubation.

Exclusion Criteria:

* known, difficult airway
* loose teeth
* pregnant
* require a rapid sequence induction,
* Body Mass Index under 30
* unable to give consent
* if special endotracheal tube (ETT) is needed for the case.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-02; Primary Completion 2009-06 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Sessler, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Comparator: Fiberoptic Intubation: Subjects will be intubated with the Fiberoptic laryngoscope.
  Active Comparator: GlideScope® Video Laryngoscope Subjects will be intubated with the GlideScope® Video Laryngoscope
Period: Overall Study
Arm/Group | Active Comparator: Fiberoptic Intubation | GlideScope® Video Laryngoscope
Started | 37 | 38
Completed | 37 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fiberoptic Intubation | GlideScope® Video Laryngoscope | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (11) | 52 (16) | 53 (13)
Gender [Count of Participants; unit: Participants]
  Female | 18 | 26 | 44
  Male | 19 | 12 | 31
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 36 | 33 | 69
  Others | 1 | 5 | 6
Region of Enrollment [Number; unit: participants]
  United States | 37 | 38 | 75
Weight [Median (Inter-Quartile Range); unit: Kg] | 117 [95 to 141] | 104 [93 to 117] | 110 [93 to 126]
Height [Mean (Standard Deviation); unit: cm] | 171 (12) | 167 (10) | 169 (11)
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 37 [33 to 49] | 36 [34 to 44] | 37 [33 to 46]
ASA physical status [Number; unit: participants]
  I: A normal healthy patient | 1 | 3 | 4
  II: A patient with mild systemic disease | 21 | 18 | 39
  III: A patient with severe systemic disease | 15 | 17 | 32
Modified Mallampati classification [Number; unit: participants] — Modified Mallampati classification was not collected for one patient in the GlideScope Video Laryngoscope group.
  participants
    I: Soft palate, uvula, fauces, pillars visible. | 7 | 8 | 15
    II: Soft palate, uvula, fauces visible. | 19 | 19 | 38
    III: Soft palate, base of uvula visible. | 10 | 8 | 18
    IV: Only hard palate visible. | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Time to Intubation (TTI) as Measured in Seconds
Description: Time from insertion of either the GlideScope or in the case of fibreoptic intubation, a Williams airway (SunMed, Largo, FL, USA) into the mouth, to the time when end-tidal PCO2 exceeded 2.7 kPa (20 mmHg).
Time Frame: from start of intubation to successfully intubated up to 100 seconds
Measure: Median (Inter-Quartile Range); unit: seconds
Groups:
- Active Comparator: Fiberoptic Intubation: Subjects will be intubated with the Fiberoptic laryngoscope.
Arm/Group | Active Comparator: Fiberoptic Intubation | GlideScope® Video Laryngoscope
Number analyzed (Participants) | 37 | 38
seconds | 43 [35 to 58] | 37 [25 to 48]
Statistical Analysis 1: Comparison: Active Comparator: Fiberoptic Intubation vs GlideScope® Video Laryngoscope; Test type: Superiority or Other; p = 0.19, Regression, Cox; Intubations accomplished with another device due to difficulty with assigned device and those took >180 s were considered as failed intubations

2. Secondary Outcome: Intubation Difficulty Score
Description: Intubation difficulty score is a 100-mm-long visual analogue scale (100 mm = extremely difficult);
Time Frame: from start of intubation to successfully intubated
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Fiberoptic Intubation | GlideScope® Video Laryngoscope
Number analyzed (Participants) | 37 | 38
units on a scale | 20 [11 to 40] | 15 [10 to 21]
Statistical Analysis 1: Comparison: Fiberoptic Intubation vs GlideScope® Video Laryngoscope; Test type: Superiority or Other; p = 0.58, ANCOVA; Ratio of Geometric Means = 0.89, 95% CI 2-sided [0.58 to 1.35] — The mean intubation difficulty score was tested after logarithmic transformation, and then back transformed for the estimated treatment effect

3. Secondary Outcome: Successful Intubation on 1st Attempt
Time Frame: from start of first intubation to end of first intubation attempt
Measure: Number; unit: participants
Arm/Group | Fiberoptic Intubation | GlideScope® Video Laryngoscope
Number analyzed (Participants) | 37 | 38
participants | 31 | 36
Statistical Analysis 1: Comparison: Fiberoptic Intubation vs GlideScope® Video Laryngoscope; Test type: Superiority or Other; p = 0.15, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.13, 95% CI 2-sided [0.95 to 1.33]

4. Secondary Outcome: Occurrence of Hypoxaemia
Description: Arterial oxygen saturation was recorded at 1 min prior to intubation, intubation, and 2, 4, 6, 8, and 10 min after; hypoxaemia was defined as occurrence of arterial oxygen saturation <90% at any of the above measurements.
Time Frame: at 1 min prior to intubation, intubation, and 2, 4, 6, 8, and 10 min after
Measure: Number; unit: participants
Arm/Group | Fiberoptic Intubation | GlideScope® Video Laryngoscope
Number analyzed (Participants) | 37 | 38
participants | 2 | 4
Statistical Analysis 1: Comparison: Fiberoptic Intubation vs GlideScope® Video Laryngoscope; Test type: Superiority or Other; p = 0.57, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.67, 95% CI 2-sided [0.28 to 10.2]

5. Secondary Outcome: Trace Bleeding
Description: Trace bleeding is a binary outcome: yes or no, which is determined based on amount of post-intubation bleeding present in the suction tube
Time Frame: Right after intubation
Measure: Number; unit: participants
Arm/Group | Fiberoptic Intubation | GlideScope® Video Laryngoscope
Number analyzed (Participants) | 37 | 38
participants | 1 | 1
Statistical Analysis 1: Comparison: Fiberoptic Intubation vs GlideScope® Video Laryngoscope; Test type: Superiority or Other; p = 0.79, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.93 to 1.09]

6. Secondary Outcome: Sore Throat Grade
Time Frame: On the first postoperative day
Population: This outcome was not collected for 1 patient in each group.
Measure: Number; unit: participants
Arm/Group | Fiberoptic Intubation | GlideScope® Video Laryngoscope
Number analyzed (Participants) | 36 | 37
participants
  None | 19 | 21
  Mild | 14 | 11
  Moderate | 2 | 3
  Severe | 1 | 2
Statistical Analysis 1: Comparison: Fiberoptic Intubation vs GlideScope® Video Laryngoscope; Test type: Superiority or Other; p = 0.82, Regression, Logistic; proportional odds logistic regression model; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.45 to 2.76]

7. Secondary Outcome: Number of Intubation Attempts
Time Frame: from start of intubation to successfully intubated
Measure: Number; unit: participants
Arm/Group | Fiberoptic Intubation | GlideScope® Video Laryngoscope
Number analyzed (Participants) | 37 | 38
participants
  1 | 31 | 36
  2 | 3 | 1
  3 | 2 | 0
  4 | 1 | 1

ADVERSE EVENTS:
Groups:
- Fiberoptic: Subjects will be intubated with the Fiberoptic laryngoscope.
Arm/Group | Fiberoptic | GlideScope® Video Laryngoscope
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/38
Other Adverse Events (participants affected / at risk) | 0/37 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes